CLINICAL TRIAL: NCT05488171
Title: Abuse Potential and Human Pharmacology of Methylone
Acronym: METI/FIS/1
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Germans Trias i Pujol Hospital (Other)
Collaborators: Fundació Recerca Institut Germans Trias i Pujol (Unknown); Istituto Superiore di Sanità (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: HUGTP/METI/FIS/1
Record Dates: First submitted 2022-02-04; First posted 2022-08-04 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Substance Use; Healthy Subjects
Keywords: methylone; pharmacokinetics; acute effects; MDMA; abuse liability; human pharmacology
MeSH Terms: conditions — Substance-Related Disorders | interventions — methylone; N-Methyl-3,4-methylenedioxyamphetamine

STUDY DESIGN:
Intervention Model Description: The protocol comprises a pilot study (n= 12) and a definitive study (n=17, 14 men and 3 women).
  The pilot study was a phase I dose-finding study that included 4 cohorts of 3 subjects (cohort 1,2,3 and 5). The conditions of each cohort were: 50 and 100 mg of methylone and placebo in cohort 1 (n= 3); 100 and 150 mg of methylone and placebo in cohort 2 (n= 3); 150 and 200 mg of methylone and placebo in cohort 3 (n= 3); 200 mg of methylone, 100 mg of MDMA and placebo in cohort 5 (n= 3). For safety reasons in cohorts 1-2-3, lower doses were allocated before the higher doses.
  After completion, the pilot study allowed defining the treatment conditions and interventions of the definitive study. The present definitive study was designed as double-blind, placebo-controlled, crossover and randomized. Each subject will participate in three experimental sessions, in each one treatment will be administered. Study treatment conditions are 200 mg of methylone, 100 mg of MDMA and placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Identical white hard gelatin capsules
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Methylone (Experimental): Methylone (3,4-methylenedioxy-N-methylcathinone) 200 mg, single dose, oral administration
  Interventions: Drug: Methylone
- 3,4-methylenedioxymethamphetamine (MDMA) (Active Comparator): MDMA (3,4-methylenedioxymethamphetamine) 100 mg, single dose, oral administration
  Interventions: Drug: 3,4-methylenedioxymethamphetamine
- Maltodextrin (Placebo Comparator): Placebo, single dose, oral administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylone — Single oral dose of 200 mg of methylone.
  Other Names: 3,4-methylenedioxy-N-methylcathinone; MDMC
  Arms: Methylone
Drug: 3,4-methylenedioxymethamphetamine — Single oral dose of 100 mg of MDMA.
  Other Names: MDMA; Ecstasy
  Arms: 3,4-methylenedioxymethamphetamine (MDMA)
Drug: Placebo — Single oral dose of placebo.
  Other Names: Non active treatment
  Arms: Maltodextrin

SUMMARY:
The purposes of the study are 1) To assess the abuse potential of methylone after controlled administration of a single oral dose of methylone 2) to evaluate subjective and physiological effects of methylone 3) to determine the pharmacokinetics parameters and metabolism of methylone.

DETAILED DESCRIPTION:
Methylone is a synthetic cathinone that has been popularized as an alternative to other illegal psychostimulants as methylenedioxymethamphetamine (MDMA, ecstasy) or mephedrone. Chemically, methylone is a beta-keto analogue of ecstasy with similar pharmacological effects in animals. To date, the available data about the human pharmacology of methylone in humans is very scarce and is mainly provided by users' experience published in internet forums or intoxication reports.

A pilot study was carried out to select the methylone dose used in this study. This current study is aimed 1) To assess the abuse potential of methylone after controlled administration of a single oral dose of methylone 2) to evaluate subjective and physiological effects of methylone 3) to determine the pharmacokinetics parameters and metabolism of methylone.

ELIGIBILITY:
Inclusion Criteria:

* Understanding and accepting all the study procedures and signing the informed consent.
* Healthy male and female volunteers aged between 18 and 45.
* Clinical history and physical examination demonstrating no organic or psychiatric disorders.
* The electrocardiogram and general blood and urine laboratory tests performed before the study must be within normal ranges. Minor or occasional changes from normal ranges are accepted if, in the investigator's opinion, considering the current state of the art, they are not clinically significant, are not life-threatening for the subjects and do not interfere with the product assessment. These changes and their non-relevance will be justified in writing specifically.
* Body weight between 50 and 90 kg and body mass index (BMI) between 19-27 kg/m². In case of women, they must weight at least 55 kg to participate. Lower or higher weights and/or BMIs will be accepted if the researchers consider that do not pose a risk to the subjects and do not interfere with the objectives of the study.
* Recreational use of methylone or other synthetic cathinones, amphetamines and/or ecstasy at least 6 occasions (two in the previous year) without serious adverse reactions.
* Women who have regular 26-32 day menstrual cycles (maximum 35 days). Participation only in follicular phase of menstrual cycle.
* Participants who agree to use reliable methods of contraception during the study such as abstinence, intrauterine devices, barrier methods with or without spermicide, or who have a vasectomized partner.

Exclusion Criteria:

* Present history of a substance use disorder according to Diagnostic and Statistical Manual for Mental Disorders (DSM-V), except for nicotine. Past history of mild substance use disorder (corresponding to substance abuse according to DSM-IV) could be included.
* Having had any somatic disease or having undergone major surgery in the 3 months prior to inclusion in the trial.
* Individual psychiatric history or schizophrenia in first-degree relatives.
* Previous or actual psychiatric disorders, alcoholism, abuse of prescription drugs or illegal substances or regular consumption of psychoactive drugs.
* Daily consumption of >40 grams of alcohol and/or >20 cigarettes.
* Blood donation 8 weeks before or participation in other clinical trials with drugs in the previous 12 weeks. In the exceptional case of having participated in this study, there is a washout period of 2 months.
* History of allergy or serious adverse reactions to medications and/or drugs.
* Pathological history or evidence of a preexisting condition (including gastrointestinal, liver, or kidney disorders) that may alter the absorption, distribution, metabolism or excretion of drugs or symptoms suggestive of drug-induced gastrointestinal irritation.
* Subjects unable to understand the nature, consequences of the study and the procedures requested to be followed.
* Subjects with positive serology to Hepatitis B, C or HIV.
* Having taken medication regularly in the month prior to the study sessions, excepting vitamins, herbal remedies or dietary supplements that, according to the researchers, do not pose a risk to the subjects and do not interfere in the objectives of the study. Single doses of symptomatic medication in the week prior to experimental sessions will be admitted if it is assumed that blood concentrations have been eliminated on the day of the experimental session.
* Women who are pregnant or breastfeeding, or who use hormonal contraceptives or do not use reliable contraceptive measures during the study (such as abstinence, intrauterine devices, barrier methods or with a vasectomized partner).
* Women with amenorrhea or severe premenstrual syndrome.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in blood pressure: Emax (peak/maximum effects) in blood pressure | Differences from baseline to 24 hours after administration
  Non-invasive systolic blood pressure (mmHg) and diastolic blood pressure (mmHg) were repeatedly recorded at baseline (45 and 30 min) prior to administration, and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10 and 24 h after administration.
  Blood pressure measured in mmHg.

SECONDARY OUTCOMES:
Change in Heart rate: Emax (peak/maximum effects) in Heart rate | Differences from baseline to 24 hours after administration
  Heart rate was repeatedly recorded at baseline (45 and 30 min) prior to administration, and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10 and 24 h after administration.
  Heart rate measured in beats per minute (bpm).
Change in Oral temperature: Emax (peak/maximum effects) in Oral temperature | Differences from baseline to 24 hours after administration
  Oral temperature was repeatedly recorded at baseline (45 and 30 min) prior to administration, and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10 and 24 h after administration.
  Oral temperature measured in Celsius degrees (ºC).
Change in Pupil diameter: Emax (peak/maximum effects) in Pupil diameter | Differences from baseline to 24 hours after administration
  Pupil diameter was repeatedly recorded at baseline (45 and 30 min) prior to administration, and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10 and 24 h after administration.
  Pupil diameter measured in millimeters (mm).
Change in Maddox Wing score (MW): Emax (peak/maximum effects) | Differences from baseline to 24 hours after administration
  Maddox wing is a device that measures the balance of extraocular muscles and quantifies exophoria as an indicator of extraocular muscle relaxation. From 22 (exophoria) to 15 (esophoria).
  It is measured at baseline (45 and 30 min) prior to administration, and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10 and 24 h.
Change in Intensity of effects: Emax (peak/maximum effects) in Intensity of effects | Differences from baseline to 24 hours after administration
  Intensity of effects will be measured using a visual analog scale (0-100 mm) at baseline (h) and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10 and 24 h after administration.
  Higher mm means more intensity of effects.
Change in High: Emax (peak/maximum effects) in High feeling | Differences from baseline to 24 hours after administration
  High will be measured using a visual analog scale (0-100 mm) at baseline and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10 and 24 h after administration.
  Higher mm means more high feeling.
Change in Stimulated: Emax (peak/maximum effects) in Stimulated feeling | Differences from baseline to 24 hours after administration
  Stimulation will be measured using a visual analog scale (0-100 mm) at baseline and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10 and 24 h after administration.
  Higher mm means more stimulation.
Change in Liking: Emax (peak/maximum effects) in Liking feeling | Differences from baseline to 24 hours after administration
  Liking will be measured using a visual analog scale (0-100 mm) at baseline and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10 and 24 h after administration.
  Higher mm means more liking.
Change in global drug effects assessed with ARCI: Emax (peak/maximum effects) in global drug effects | Differences from baseline to 24 hours after administration
  Global drug effects will be measured using the short form (49 items) of the Addiction Research Center Inventory (ARCI). This is a true/false response questionnaire with 49 items. The global results include five subscales (sedation, euphoria, dysphoria, intellectual efficiency and amphetamine-like effects.
  It is administered at baseline and 1, 2, 3, 4, 6, 8, and 10 h after administration.
  Scores range usually from a total of 12 to 57 points. More points mean more effects.
Change in global drug effects assessed with VESSPA: Emax (peak/maximum effects) in global drug effects | Differences from baseline to 24 hours after administration
  Global drug effects will be measured using the Evaluation of the Subjective Effects of Substances with Abuse Potential questionnaire (VESSPA-SSE). This questionnaire consists of 36 items (0-4 score) that evaluate subjective effects related to stimulants such as MDMA. VESSPA includes six subscales (sedation, psychosomatic anxiety, changes in perception, pleasure and sociability, activity and energy, and psychotic symptoms). Scores of each subscale ranges from 0 to 24 (maximal effects)
  It is administered at baseline and 1, 2, 3, 4, 6, 8, and 10 h after administration.
Maximum plasma concentration (Cmax) of methylone | From baseline to 24 hours after methylone administration
  Calculation of maximum concentration of methylone (ng/mL) in samples collected from 15 min prior to administration (time 0) and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10 and 24 hours.
Maximum plasma concentration (Cmax) of MDMA | From baseline to 24 hours after MDMA administration
  Calculation of maximum concentration of MDMA (ng/mL) in samples collected from 15 min prior to administration (time 0) and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10 and 24 hours.
Time to reach maximum plasma concentration (Tmax) of methylone | From baseline to 24 hours after methylone administration
  Time (h) to reach maximum concentration of methylone in plasma after administration.
Time to reach maximum plasma concentration (Tmax) of MDMA | From baseline to 24 hours after MDMA administration
  Time (h) to reach maximum concentration of MDMA in plasma after administration.
Area under the concentration-time curve (AUC 0-24 h) of methylone in plasma concentrations | From baseline to 24 hours after methylone administration
  Calculation of AUC with samples collected from 15 min prior (time 0) and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10 and 24 hours after methylone administration.
Area under the concentration-time curve (AUC 0-24 h) of MDMA in plasma concentrations | From baseline to 24 hours after MDMA administration
  Calculation of AUC with samples collected from 15 min prior (time 0) and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10 and 24 hours after MDMA administration.
Maximum oral fluid concentration (Cmax) of methylone | From baseline to 24 hours after methylone administration
  Calculation of maximum concentration (ng/mL) of methylone in oral fluid (saliva) samples collected with a Salivette device at the same time points as serum. Oral fluid is collected 15 min before administration (time 0), at to 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10 and 24 hours.
Maximum oral fluid concentration (Cmax) of MDMA | From baseline to 24 hours after MDMA administration
  Calculation of maximum concentration (ng/mL) of MDMA in oral fluid (saliva) samples collected with a Salivette device at the same time points as serum. Oral fluid is collected 15 min before administration (time 0), at to 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10 and 24 hours.
Time to reach maximum oral fluid concentration (Tmax) of methylone | From baseline to 24 hours after methylone administration
  Time (h) to reach maximum concentration of methylone in oral fluid after administration.
Time to reach maximum oral fluid concentration (Tmax) of MDMA | From baseline to 24 hours after MDMA administration
  Time (h) to reach maximum concentration of MDMA in oral fluid after administration.
Area under the concentration-time curve (AUC 0-24h) of methylone oral fluid concentrations | From baseline to 24 hours after methylone administration
  Calculation of AUC with oral fluid samples collected from 15 min prior to methylone administration (time 0) and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10 and 24 hours.
Area under the concentration-time curve (AUC 0-24h) of MDMA oral fluid concentrations | From baseline to 24 hours after MDMA administration
  Calculation of AUC with oral fluid samples collected from 15 min prior to MDMA administration (time 0) and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10 and 24 hours.
Total amount methylone excreted in 24 h urine samples. | From baseline to 24 hours after methylone administration
  Urine was collected 15 minutes before administration (time 0) and then between 0-4 h, 4-8 h, 8-12 h, and 12-24 h after methylone administration.
Total amount MDMA excreted in 24 h urine samples. | From baseline to 24 hours after MDMA administration
  Urine was collected 15 minutes before administration (time 0) and then between 0-4 h, 4-8 h, 8-12 h, and 12-24 h after MDMA administration.
Total concentration of methylone present in sweat | From baseline to 12 hours after methylone administration
  Concentration of methylone in ng/patch. Samples were collected with dermal patches (5 x 5 cm areas) applied to the back and removed at different intervals such as: 0-2 h, 0-4 h, 0-6 h, 0-8 h, and 0-10 h, 10-12 h.
Total concentration of MDMA present in sweat | From baseline to 12 hours after MDMA administration
  Concentration of MDMA in ng/patch. Samples were collected with dermal patches (5 x 5 cm areas) applied to the back and removed at different intervals such as: 0-2 h, 0-4 h, 0-6 h, 0-8 h, and 0-10 h, 10-12 h.
Pharmacological class identification | Only administered 8 hours after administration
  In the pharmacological class identification questionnaire, the participant selects the pharmacological class that better describes the administered drug.
  This questionnaire is administered 8 h after administration.
Change in psychomotor vigilance task (PVT): Emax (peak/maximum effects) | Differences from baseline to 2 hours after administration
  Test will be performed using specific computer software that assesses simple reaction time to a numeric stimulus. Results are milliseconds (increased simple reaction time is related to worst psychomotor performance) It is measured at baseline (45 and 30 min) prior to administration, and at 1 and 2 h.
Psychiatric evaluation using Young Mania Rating Scale (YMRS) | Differences from baseline to 6 hours after administration
  YMRS (11 items) assessing manic symptoms from 0 to 4 (total score from 0 to 44).
  It is measured at baseline (30 min) prior to administration, and at 0.5, 1, 4, and 6 h after administration.
  A higher score indicates a higher severity of mania.

CONTACTS AND LOCATIONS:
Overall Officials: Magi Farré, MD, PhD, Principal Investigator — Germans Trias i Pujol Hospital
Locations (1):
- Germans Trias i Pujol Hospital, Badalona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Poyatos L, Perez-Mana C, Hladun O, Nunez-Montero M, de la Rosa G, Martin S, Barriocanal AM, Carabias L, Kelmendi B, Taoussi O, Busardo FP, Fonseca F, Torrens M, Pichini S, Farre M, Papaseit E. Pharmacological effects of methylone and MDMA in humans. Front Pharmacol. 2023 Feb 17;14:1122861. doi: 10.3389/fphar.2023.1122861. eCollection 2023. PMID 36873994